CLINICAL TRIAL: NCT01393002
Title: Web-based Structured Survey of Retrospective Data of Invasive Mycosis in Intensive Care Patients in Berlin - Brandenburg
Brief Title: Perception and Prevalence of Fungal Infections in Berlin - Brandenburg
Acronym: IFI_ICU
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Claudia Spies, Department of Anesthesiology and Intensive Care Medicine CVK/CCM, Charite University, Berlin, Charite University, Berlin, Germany
Other Study IDs: IFI_ICU
Record Dates: First submitted 2011-07-05; First posted 2011-07-13 (Estimated); Last update posted 2013-10-18 (Estimated); Status verified 2013-10

CONDITIONS: Invasive Mycosis
Keywords: intensive care; candidemia; fungal infection
MeSH Terms: conditions — Invasive Fungal Infections; Candidemia; Mycoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- INABBRA: Participating hospitals in the INABBRA alliance.

SUMMARY:
This is a structured web-based survey in selected hospitals with intensive care units in Berlin- Brandenburg that will focus on the analysis of current knowledge in ICUs in the field of invasive mycoses.

DETAILED DESCRIPTION:
Intensive care patients with invasive mycosis require a special clinical expertise especially in light of a high lethality. Early identification of patients at risk to develop a fungal infection is of utmost importance to start effective antifungal therapy. The implementation of current knowledge into clinical practice to fight fungal infection is not clear.

ELIGIBILITY:
Inclusion Criteria:

* Intensive care units of hospitals in the INABBRA alliance.
* Patients with invasive mycosis.

Exclusion Criteria:

* Hospitals without intensive care unit.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Intensive care units of different primary and secondary care hospitals in the region of Berlin-Brandenburg.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Perception and prevalence of fungal infections | 4 months
  Perception and prevalence of fungal infections in ICU patients differs from real prevalence and leads to insufficient attribution of importance to this special medical condition.

SECONDARY OUTCOMES:
Practice - Surrogate markers for diagnosis and therapy of fungal infection and retrospective analysis of cases of invasive mycosis in a peer-review setting. | 6 months
  Qualitative and quantitative estimation of surrogate markers for diagnosis and treatment of invasive mycosis
  Number of bloodcultures per year Rate of bloodcultures positive for fungi ICD-10 diagnosis ICU length of stay for patients with invasive mycosis and/or fungal infection Hospital mortality for patients with invasive mycosis and/or fungal infection Number of patients treated by antimycotics per year Mean duration of antifungal treatment Defined daily doses of antimycotics given by hospital pharmacy

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Spies, Prof., MD, Study Director — Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Virchow-Klinikum and Campus Charité Mitte, Charité - Universitaetsmedizin Berlin, Berlin, State of Berlin, Germany

REFERENCES:
- [Background] Morrell M, Fraser VJ, Kollef MH. Delaying the empiric treatment of candida bloodstream infection until positive blood culture results are obtained: a potential risk factor for hospital mortality. Antimicrob Agents Chemother. 2005 Sep;49(9):3640-5. doi: 10.1128/AAC.49.9.3640-3645.2005. PMID 16127033